CLINICAL TRIAL: NCT02296645
Title: A Pilot Clinical Evaluation of the Antimicrobial Effectiveness of Topically Applied ZuraPrep™
Brief Title: Efficacy Study to Evaluate Antimicrobial Effectiveness of ZuraPrep™ (ZX-ZP-0055)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ZX-ZP-0055 (MBT# 865-101)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2015-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — citrate, isopropyl alcohol, methylene blue, parabens drug combination; Ethanol; Chromogranins; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZuraPrep (Experimental): Isopropyl alcohol (IPA) (70%)
  Interventions: Drug: ZuraPrep
- ChloraPrep (Active Comparator): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ChloraPrep

INTERVENTIONS:
Drug: ZuraPrep — Apply topically.
  Other Names: Isopropyl alcohol 70%
  Arms: ZuraPrep
Drug: ChloraPrep — Apply topically.
  Other Names: CHG 2% / IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: ChloraPrep

SUMMARY:
This is a randomized, paired-comparisons design where each subject receives two of the planned treatments.

DETAILED DESCRIPTION:
ZuraPrep is being evaluated for safety and efficacy as a preoperative skin preparation against the Tentative Final Monograph (TFM) 10-minute end point recently revised by the FDA for the lower bound of a 95% confidence interval whereas there must be specific reductions of normal flora in the abdomen and groin areas. A positive control will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Subjects to whom all of these conditions apply will be eligible for enrollment in this study:

  * Males and/or females, at least 18 years or older. Are in good general health.
  * Have skin within 6 inches of the test sites that is free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders.
  * Cooperative and willing to follow Subject Instructions (Appendix 14.6).
  * Cooperative and willing to sign Consent Form and HIPAA Authorization Form.
  * Have Screening Day baseline counts of at least 1.3 x 103 CFU/cm2 per abdominal site (left and right) and 1.0 x 105 CFU/cm2 per groin site (left and right). For replacement subjects, have Screening Day baseline counts of at least 1.3 x 103 CFU/cm2 per abdominal site (left and right) and/or 1.0 x 105 CFU/cm2 per groin site (left and right).

Exclusion Criteria:

* Subjects to whom any of these conditions apply will be excluded from this study:

  * Topical or systemic antimicrobial exposure within 14 days prior to Screening Day. Restrictions include, but are not limited to antimicrobial soaps, antiperspirants/deodorants, shampoos, lotions, perfumes, after shaves, colognes, and topical or systemic antibiotics.
  * Swimming in chemically treated pools or bathing in hot tubs, spas and whirlpools within 14 days prior to Screening Day.
  * Use of tanning beds, hot waxes, or depilatories, including shaving (in the applicable test areas) within 14 days prior to Screening Day.
  * Contact with solvents, acids, bases, fabric softener-treated clothing or other household chemicals in the applicable test areas within 14 days of the Screening Day. Subjects who have a history of sensitivity to natural rubber latex, adhesive skin products (e.g., Band-Aids, medical tapes), isopropyl alcohol, citric acid, methylene blue, methylparaben, propylparaben, or chlorhexidine gluconate chlorhexidine gluconate products.
  * Subjects who have a history of diabetes.
  * Subjects who have a history of skin allergies.
  * Subjects who have a history of skin cancer within 6 inches of the applicable test areas.
  * Subjects who are pregnant, attempting pregnancy or nursing.
  * Subjects who have showered or bathed within 48 hours of the Screening Day or Treatment Day (sponge baths may be taken, however, the lower abdomen and upper thigh region must be avoided).
  * Subjects who receive an irritation score of 1 for any individual skin condition prior to the Screening Day baseline or Treatment Day baseline sample collection.
  * Participation in another clinical trial in the 30 days prior to Test Day of this study (treatment with test materials in this study), or be currently enrolled in another clinical trial, or has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Reduction of skin flora | 10 minutes
  The primary measure of antimicrobial efficacy is the log10 reduction of skin flora on the abdominal and groin sites 10 minutes following application of the study treatments relative to the Treatment Day baseline log10 counts.

CONTACTS AND LOCATIONS:
Overall Officials: M. Hamid Bashir, MD, Principal Investigator — MicroBioTest, Division of Microbac Laboratories, Inc.
Locations (1):
- MicroBioTest Laboratories, Sterling, Virginia, United States